CLINICAL TRIAL: NCT07351617
Title: Translation, Validity, and Reliability of the Turkish Version of the Pain Metacognitions Questionnaire
Brief Title: Turkish Version of the Pain Metacognitions Questionnaire
Status: Not yet recruiting | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Mahmut Sürmeli, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: CKU-PMQ-TR-2025
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Pain Metacognitions
Keywords: chronic pain; pain metacognitions; questionnaire validation; reliability
MeSH Terms: conditions — Chronic Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Chronic Pain: Adults aged 18 years and older with chronic non-cancer pain who participate voluntarily in this observational study.
  Interventions: Other: No Intervention (Observational Study)

INTERVENTIONS:
Other: No Intervention (Observational Study) — This is an observational study. No intervention is administered. Data are collected using self-report questionnaires only.

SUMMARY:
Pain-related thoughts and beliefs play an important role in how individuals experience and cope with chronic pain. Metacognitions about pain, such as beliefs about the uncontrollability or harmfulness of pain-related thoughts, may influence emotional distress and pain-related outcomes. The Pain Metacognitions Questionnaire was developed to assess these beliefs; however, a validated Turkish version is not currently available. The aim of this study is to translate the Pain Metacognitions Questionnaire into Turkish and to evaluate its validity and reliability in adults with chronic non-cancer pain. This observational study will include adult individuals experiencing chronic pain for at least three months. Data will be collected using self-report questionnaires administered in a single assessment session. The findings of this study are expected to provide a reliable and valid measurement tool for assessing pain-related metacognitions in Turkish-speaking populations and to support future clinical and research applications in chronic pain management.

DETAILED DESCRIPTION:
Chronic pain is a complex condition influenced not only by biological factors but also by cognitive and emotional processes. Metacognitions, defined as beliefs about one's own thoughts, have been shown to play a significant role in the persistence and management of chronic pain. The Pain Metacognitions Questionnaire was developed to assess pain-related metacognitive beliefs, including perceptions about the uncontrollability, danger, and usefulness of pain-related thoughts. Despite its growing use in research, a validated Turkish version of this questionnaire is currently lacking.

This study is designed as an observational, cross-sectional investigation aiming to translate the Pain Metacognitions Questionnaire into Turkish and to examine its psychometric properties in adults with chronic non-cancer pain. The translation process will follow standard forward-backward translation procedures to ensure linguistic and conceptual equivalence. Content validity will be evaluated by expert review.

Participants will be adults aged 18 years and older who have experienced chronic non-cancer pain for at least three months. After providing informed consent, participants will complete the Turkish version of the Pain Metacognitions Questionnaire along with additional validated self-report measures assessing pain-related and psychological constructs. Data collection will be conducted through face-to-face or online survey methods, and all assessments will be completed at a single time point.

Psychometric analyses will include evaluation of internal consistency, test-retest reliability, construct validity, and factor structure. Correlational analyses will be used to examine relationships between pain metacognitions and related psychological variables. The results of this study are expected to contribute to the assessment of cognitive processes in chronic pain and to provide a valid and reliable instrument for use in Turkish clinical and research settings.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Experiencing chronic non-cancer pain for at least three months
* Ability to read and understand Turkish
* Voluntary participation and provision of informed consent

Exclusion Criteria:

* Presence of cancer-related pain
* Severe cognitive impairment preventing completion of questionnaires
* Incomplete or incorrectly completed questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 years and older with chronic non-cancer pain.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-19 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Pain Metacognitions Score | At enrollment (single assessment)
  Pain metacognitions will be assessed using the Turkish version of the Pain Metacognitions Questionnaire. The questionnaire evaluates metacognitive beliefs related to pain, including beliefs about the uncontrollability, danger, and usefulness of pain-related thoughts. Higher scores indicate more maladaptive pain-related metacognitions.

SECONDARY OUTCOMES:
Pain Intensity | At enrollment (single assessment)
  Pain intensity will be measured using a numerical rating scale as part of the Brief Pain Inventory, where higher scores indicate greater pain intensity.
Pain Interference | At enrollment (single assessment)
  Pain interference will be assessed using the Brief Pain Inventory, evaluating the extent to which pain interferes with daily activities and functioning. Higher scores indicate greater pain-related interference.
Pain Catastrophizing | At enrollment (single assessment)
  Pain catastrophizing will be measured using a validated self-report questionnaire assessing rumination, magnification, and helplessness related to pain. Higher scores indicate greater levels of pain catastrophizing.
Anxiety and Depression Symptoms | At enrollment (single assessment)
  Symptoms of anxiety and depression will be evaluated using a validated self-report scale. Higher scores indicate greater psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin University, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality considerations.